CLINICAL TRIAL: NCT04604080
Title: Post-COVID-19 Epidemic Depression Assessment in Adults in South Punjab Pakistan
Status: Completed | Type: Observational
Sponsor: Islamia University of Bahawalpur (Other)
Responsible Party: Principal Investigator, Jafir Hussain Shirazi, Lecturer, Islamia University of Bahawalpur
Other Study IDs: U1111-1260-1614
Record Dates: First submitted 2020-10-25; First posted 2020-10-27 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Depression, Anxiety
Keywords: Depression; Anxiety; Epidemiology
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single group: Respondents will be given survey form, filled and will be collected back
  Interventions: Other: service of questionnaire

INTERVENTIONS:
Other: service of questionnaire — Respondents will be given a survey form only and after filling this will be collected back

SUMMARY:
To assess the depression in adults especially in post COVID-19 duration in the rural and urban settings.

DETAILED DESCRIPTION:
This study is designed to assess the prevalence of depression after the general and smart lockdown in various areas. This study includes both genders of any age.

ELIGIBILITY:
Inclusion Criteria:Any individual who can respond to the given questionnaire, with or without any ailment will be included in this study -

Exclusion Criteria:

Unconcious and non-cooperative individuals

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents/ Visitors of the south punjab will be the study population of this study
Sampling Method: Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Prevalence estimation of depression in adults | study will be completed in 15 days maximum
  % prevalence of depression in adult population of south punjab will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Jafir Shirazi, PhD, Principal Investigator — The Islamia University of Bahawalpur
Locations (5):
- Pakistan (5):
  - The Islamia University of Bahawalpur, Chak Four Hundred Fifty-four, Punjab Province
  - GC University Faisalabad, Faisalabad, Punjab Province
  - University of Veterinary and Animal Sciences, Lahore, Lahore, Punjab Province
  - Bahauddin Zakriya University Multan, Multan, Punjab Province
  - Quaid-i-Azam University Islamabad, Islamabad

IPD SHARING:
Plan to Share IPD: No